CLINICAL TRIAL: NCT00395824
Title: Heparin-Coated Polyacrylonitrile Membrane Versus Regional Citrate Anticoagulation: a Prospective Randomised Study of 2 Anticoagulation Strategies in Patients at Risk of Bleeding
Brief Title: Citrate Anticoagulation vs. Heparin-Coated Dialyzers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pe2006-01
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Dialysis
Keywords: citrate; anticoagulation; heparin-coated membrane

INTERVENTIONS:
Procedure: anticoagulation procedure

SUMMARY:
Hemodialysis causes contact activation of the coagulation pathway (1). For this reason, unfractionated or low molecular weight heparins are administered in daily practice to prevent thrombosis of the dialyzer and blood circuit, but the dose commonly used causes systemic anticoagulation. This can cause serious complications in patients with high risk of bleeding. Regional and low-dose heparinization, use of prostacycline, regional citrate anticoagulation (RCA), and high-flow-rate hemodialysis without anticoagulation have been shown to reduce bleeding complications. Each of these methods, however, is characterized by its own technical difficulties, limitations, or complications.

The present study aimed to compare the efficacy and safety of heparin-coated polyacrylonitrile membranes (AN69ST) and regional citrate anticoagulation in hemodialysis patients at risk of bleeding

DETAILED DESCRIPTION:
1. Open label single centre prospective randomized trial including 33 patients aged over 18 years with chronic kidney disease stage 5 requiring intermittent hemodialysis at the University Hospital Leuven and at risk of bleeding. Exclusion criteria were: any haemostatic disorder favouring either bleeding or clotting, anti-vitamin K or heparin treatment, heparin induced thrombocytopenia and haemodynamic instability. Written informed consent before enrolment.
2. Random allocation (by sealed enveloppe) to RCA with a calcium free dialysate (RCA-Ca0), RCA with a calcium containing dialysate (RCA-Ca1,5) or to anticoagulant-free hemodiaysis with a heparin-coated polyacrylonitrile membrane (Nephral 300ST®).
3. At the end of each dialysis session, arterial and venous drip chambers and the filter will be inspected for visible signs of coagulation. Corresponding to the standard care at our dialysis unit, a semi-quantitative score with a range from 0 (no signs of clotting) to 4 (complete occlusion) will be used for evaluation of the dialyzer. By definition, the drip chamber will be considered clotted when a thrombus was visible after the rinse back procedure. A fibrin ring against the wall of the drip chamber will be considered normal.
4. Blood samples for assessment of prothrombin fragment F1+2 and d-dimers will be collected from the inlet blood catheter prior to hemodialysis initiation and during hemodialysis at T15, T120 and T238.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* chronic kidney disease stage 5 requiring intermittent hemodialysis
* at risk of bleeding
* written informed consent

Exclusion Criteria:

* any haemostatic disorder favouring either bleeding or clotting
* anti-vitamin K or heparin treatment
* heparin induced thrombocytopenia
* haemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33
Dates: Start 2005-01; Study Completion 2005-09

PRIMARY OUTCOMES:
anticoagulation efficacy as evaluated by clotting score of dialyser
anticoagulation efficacy as evaluated by occurrence of major and minor clotting events
anticoagulation efficacy as evaluated by instantaneous blood clearances

SECONDARY OUTCOMES:
anticoagulation efficay as evaluated by time course of coagulation parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hopsital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Evenepoel P, Dejagere T, Verhamme P, Claes K, Kuypers D, Bammens B, Vanrenterghem Y. Heparin-coated polyacrylonitrile membrane versus regional citrate anticoagulation: a prospective randomized study of 2 anticoagulation strategies in patients at risk of bleeding. Am J Kidney Dis. 2007 May;49(5):642-9. doi: 10.1053/j.ajkd.2007.02.001. PMID 17472846